CLINICAL TRIAL: NCT06553560
Title: Investigation of the Postoperative Analgesic Effect of the Combination of Superficial Parasternal Block (PSB) and Recto-Intercostal(İC) Fascial Plane Block in Patients Undergoing Cardiac Surgery Via Sternotomy: Case Series
Brief Title: The Efficacy of PSB and Recto-intercostal Block Combination on Postoperative Pain in Patients Undergoing Cardiac Surgery Via Sternotomy: Case Series
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Associate Professor, Cumhuriyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PSB and Recto-İC in sternotomy
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Post Operative Pain
Keywords: sternotomy; cardiac surgery; parasternal block; recto-intercostal fascial plane block; postoperative pain; regional anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parasternal Block and Recto-İntercostal Fascial Plane Block (Other): Superficial PSB is performed with the patient in the supine position using a high-frequency linear USG probe. The probe is placed longitudinally 2 cm lateral to the sternal border to visualize the T2-T4 intercostal space and to identify the pectoralis major muscle, intercostal muscle, and pleura. 10 ml of 0.25% bupivacaine local anesthetic is administered between the pectoralis major and intercostal muscle using an in-plane approach with a 100 mm needle. In addition, a Recto-Intercostal Fascial Plane Block is performed with a high-frequency linear USG probe. The probe is placed 2-3 cm lateral to the xiphoid so that the rectus abdominis muscle and 6-7th cartilages are visualized. The needle is advanced to the plane between the costal cartilage and the rectus abdominis muscle using the in-plane technique and 1-2 ml of saline is injected. After observing the spread to the target plane, 20 ml of 0.25% bupivacaine is applied. The same process is repeated bilaterally.
  Interventions: Other: Parasternal Block and Recto-İntercostal Fascial Plane Block

INTERVENTIONS:
Other: Parasternal Block and Recto-İntercostal Fascial Plane Block — Superficial PSB is performed with the patient in the supine position using a high-frequency linear USG probe. The probe is placed longitudinally 2 cm lateral to the sternal border to visualize the T2-T4 intercostal space and to identify the pectoralis major muscle, intercostal muscle, and pleura. 10 ml of 0.25% bupivacaine local anesthetic is administered between the pectoralis major and intercostal muscle using an in-plane approach with a 100 mm needle. In addition, a Recto-Intercostal Fascial Plane Block is performed with a high-frequency linear USG probe. The probe is placed 2-3 cm lateral to the xiphoid so that the rectus abdominis muscle and 6-7th cartilages are visualized. The needle is advanced to the plane between the costal cartilage and the rectus abdominis muscle using the in-plane technique and 1-2 ml of saline is injected. After observing the spread to the target plane, 20 ml of 0.25% bupivacaine is applied. The same process is repeated bilaterally.

SUMMARY:
The aim of this study was to investigate the effectiveness of the combination of Superficial Parasternal Block and Recto-Intercostal Fascial Plane Block in patient groups undergoing cardiac surgery via sternotomy by evaluating postoperative pain scores and analgesic consumption.

DETAILED DESCRIPTION:
Ten patients received a combination of parasternal block and recto-intercostal fascial plane block as an intervention. Patients received bilateral parasternal block and recto-intercostal fascial plane block with 0.25% bupivacaine (total volume 60 ml) in the operating room before surgery. All blocks will be performed after general anesthesia induction, before skin incision. All patients included in the study will be given 50 mg dexketoprofen and 1 g paracetamol intravenously (i.v.) 10 minutes before skin closure. All patients will be given 3x1 g iv paracetamol and 2x50 mg dexketoprofen within the first 24 hours postoperatively. Numerical rating scale (NRS) was used to assess pain at the 1st, 6th, 12th, 18th and 24th hours after surgery. Total morphine consumption was calculated using a patient-controlled analgesia (PCA) device. Tramadol was planned as rescue analgesic medication (maximum dose: 300 mg/day).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age who will undergo cardiac surgery with sternotomy under general anesthesia and who are in classes I-II-III according to the American Society of Anesthesiologists (ASA) risk classification.

Exclusion Criteria:

* Patients who did not give consent,

  * patients with coagulopathy,
  * patients with signs of infection at the block application site,
  * patients using anticoagulants,
  * patients with local anesthetic drug allergies,
  * patients with unstable hemodynamics,
  * patients who could not cooperate during postoperative pain assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Comparing the numerical rating scale scores | Postoperative 24 hours
  Numerical rating scale will be used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Comparing total morphine consumption | Postoperative 24 hours
  Postoperative analgesic need

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Gündoğdu, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation